CLINICAL TRIAL: NCT03436030
Title: Atrial and Ventricular Wall Stress, Effects of Breathing and Airway Pressure
Brief Title: Atrial and Ventricular Wall Stress During Breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-327-31M
Record Dates: First submitted 2017-12-15; First posted 2018-02-19 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2018-02

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Healthy reclining adult volunteers, with Valsalva manoeuver, Muller manoeuver, light continuous positive airway pressure by mask, passive leg raising, and maximal hand-grip. Ultrasound heart images captured before and during.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm, breathing manuevers (Experimental): All subjects perform/undergo Valsalva, Muller, CPAP, hand grip, and passive leg raise, with ultrasound examination of heart recorded before and during the manoeuvre.
  Interventions: Other: Simple breathing manuevers during brief echocardiographic imaging

INTERVENTIONS:
Other: Simple breathing manuevers during brief echocardiographic imaging — Valsalva, Muller, light mask CPAP, leg raising, hand grip.

SUMMARY:
Healthy reclining adult volunteers, with Valsalva manoeuver, Muller manoeuver, light continuous positive airway pressure by mask, passive leg raising, and maximal hand-grip. Ultrasound heart images captured before and during.

DETAILED DESCRIPTION:
With focus on atrial wall strain and strain-rate, In healthy volunteer adult subjects, heart ultrasound is recorded during resting, Valsalva manoeuver, Muller manoeuver, passive leg raising, and handgrip. Echocardiographic recordings are made before and during each intervention. Participants are otherwise resting in a reclined position.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults

Exclusion Criteria:

* known heart or lung disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-18 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in atrial wall stress during breathing manoeuver, compared to control measurement immediately before the breathing manoeuver | 30 seconds, i.e. control measurement and then measurement during breathing manoeuver observed from same breathing/measurement sequence
  Echocardiographic measure, comparing control measurement to measurement during breathing manoeuver

CONTACTS AND LOCATIONS:
Locations (1):
- Umeå University, and the University Hospital of Umeå, Umeå, Sweden

REFERENCES:
- [Derived] Gottfridsson P, A'Roch R, Lindqvist P, Law L, Myrberg T, Hultin M, A'Roch A, Haney M. Left atrial contraction strain and controlled preload alterations, a study in healthy individuals. Cardiovasc Ultrasound. 2022 Mar 30;20(1):8. doi: 10.1186/s12947-022-00278-1. PMID 35354482